CLINICAL TRIAL: NCT00680238
Title: Pregnancy and Implantation Rates When Embryos Are Selected Based on a Single Day 3 Score (Day 3)vs Graduated Embryo Score(GES) Plus Soluble Human Leukocyte Antigen-G Expression.
Brief Title: Pregnancy/Implantation Rates Using a Day 3 Score Versus Graduated Embryo Score Plus a Biochemical Marker (sHLA-G)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Responsible Party: Mr DJ Kotze, Stellenbosch University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DKotze
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Infertility
Keywords: Pregnancy; implantation; miscarriage; sHLA-G
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Urofollitropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Embryo selection for transfer based on a Day 3 score only.
  Interventions: Drug: Human derived FSH
- B (Active Comparator): Embryos for transfer by first selecting any embryos that had a positive sHLA-G expression of OD = 190 ±6 and correlating such with the highest GES score available.
  Interventions: Drug: Human derived FSH

INTERVENTIONS:
Drug: Human derived FSH — Customized for each patient
  Other Names: Bravelle

SUMMARY:
Objective: To compare pregnancy rates and implantation rates when embryos are selected based on a single Day 3 (D.3) score vs. a GES score plus sHLA-G expression.

DETAILED DESCRIPTION:
Comparing pregnancy rates and implantation rates when embryos are selected using the most common criteria for embryo selection on day 3 - the morphology-(number of blastomere, their shape and size and the percentage of fragmentation)vs a graduated embryo score accumulated over 72 hours and the expression of sHLA-G at 44-46 hours post fertilization.

ELIGIBILITY:
Inclusion Criteria:

* Self paying ART patients

Exclusion Criteria:

* Abnormal uterus
* Specific Immunologic factors

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy and implantation rates | 12 weeks

SECONDARY OUTCOMES:
Miscarriage rates | 9 months
Miscarriage rates | 9-11 day until βhCG

CONTACTS AND LOCATIONS:
Overall Officials: Thinus Kruger, M.D. PhD., Study Director — University of Stellenbosch